CLINICAL TRIAL: NCT05113745
Title: A Study to Assess the Long-term Efficacy and Safety of AXS-12 in the Treatment of Cataplexy and Excessive Daytime Sleepiness in Subjects With Narcolepsy
Brief Title: A Study to Assess the Long-term Efficacy and Safety of AXS-12 (Reboxetine) in Subjects With Narcolepsy (ENCORE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AXS-12-302
Record Dates: First submitted 2021-10-29; First posted 2021-11-09 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Narcolepsy; Cataplexy; Excessive Daytime Sleepiness
Keywords: AXS-12; Narcolepsy; Cataplexy; Excessive Daytime Sleepiness; Reboxetine; Axsome
MeSH Terms: conditions — Narcolepsy; Cataplexy; Disorders of Excessive Somnolence | interventions — Reboxetine

STUDY DESIGN:
Intervention Model Description: Open-label treatment period, followed by a double-blind treatment period.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AXS-12 (reboxetine) (Experimental): * Up to 24 weeks in open-label period
  * Up to 4 weeks in randomized double-blind period
  Interventions: Drug: AXS-12 (reboxetine)
- Placebo (Placebo Comparator): Up to 4 weeks in randomized double-blind period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AXS-12 (reboxetine) — AXS-12 tablets, taken twice daily
  Arms: AXS-12 (reboxetine)
Drug: Placebo — Placebo tablets, taken twice daily
  Arms: Placebo

SUMMARY:
This study will evaluate the long-term efficacy and safety of AXS-12 in narcoleptic subjects with cataplexy and excessive daytime sleepiness (EDS).

DETAILED DESCRIPTION:
This study is a multi-center trial consisting of a 24-week open-label period, followed by a 4-week double-blind, placebo-controlled, randomized withdrawal period. At the Week 24 visit, subjects will be randomized in a 1:1 ratio either to continue to receive AXS-12 or to switch to placebo, for the next 4 weeks. Eligible subjects will have previously participated in the AXS-12-301 study.

ELIGIBILITY:
Inclusion Criteria:

* Completed the treatment period of Study AXS-12-301
* Willing and able to comply with the study requirements

Exclusion Criteria:

* Significant change in medical history or concomitant medications since enrolling in the AXS-12-301 study which, in the opinion of the Investigator, would render the subject unsuitable to receive AXS-12

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Long-term safety as measured by the incidence of treatment-emergent adverse events | Up to 28 weeks
Efficacy as measured by change in frequency of cataplexy attacks from baseline. | Baseline to Week 27

CONTACTS AND LOCATIONS:
Locations (24):
- United States (23):
  - Clinical Research Site, Phoenix, Arizona
  - Clinical Research Site, Boulder, Colorado
  - Clinical Research Site, Colorado Springs, Colorado
  - Clinical Research Site, Brandon, Florida
  - Clinical Research Site, Clearwater, Florida
  - Clinical Research Site, Doral, Florida
  - Clinical Research Site, Miami Lakes, Florida
  - Clinical Research Site, Winter Park, Florida
  - Clinical Research Site, Atlanta, Georgia
  - Clinical Research Site, Stockbridge, Georgia
  - Clinical Research Site, Chevy Chase, Maryland
  - Clinical Research Site, Kalamazoo, Michigan
  - Clinical Research Site, Novi, Michigan
  - Clinical Research Site, Neptune City, New Jersey
  - Clinical Research Site, Denver, North Carolina
  - Clinical Research Site, Gastonia, North Carolina
  - Clinical Research Site, Huntersville, North Carolina
  - Clinical Research Site, Cincinnati, Ohio
  - Clinical Research Site, Wyomissing, Pennsylvania
  - Clinical Research Site, Charleston, South Carolina
  - Clinical Research Site, Columbia, South Carolina
  - Clinical Research Site, Austin, Texas
  - Clinical Research Site, San Antonio, Texas
- Clinical Research Site, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Axsome Therapeutics Website — http://www.axsome.com